CLINICAL TRIAL: NCT06129890
Title: Neuromodulation in Patients With Neuropathic Pain and Depression: a Cross-over Study Between Two Targets in Transcranial Magnetic Stimulation, the Primary Motor Cortex and the Dorsolateral Prefrontal Cortex.
Brief Title: Neuromodulation in Patients With Neuropathic Pain and Depression.
Acronym: DOLODEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 23CH155; ANSM (Other: 2023-A01346-39)
Record Dates: First submitted 2023-10-24; First posted 2023-11-13 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Neuropathic Pain; Depression
Keywords: Neuropathic pain; Depressive Disorder; transcranial magnetic stimulation; neuromodulation; pain relief
MeSH Terms: conditions — Neuralgia; Depression; Depressive Disorder | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- M1 - DLPFC (Other): Initial primary motor cortex stimulation (M1) followed by cortex prefrontal cortex (DLPFC) :
  rTMS of M1, washout, rTMS of DLPFC
  Interventions: Device: Repetitive transcranial magnetic stimulation (rTMS) - M1/DLPFC
- DLPFC - M1 (Other): Initial cortex prefrontal cortex (DLPFC) stimulation followed by primary motor cortex stimulation (M1) :
  rTMS of DLPFC, washout, rTMS of M1
  Interventions: Device: Repetitive transcranial magnetic stimulation (rTMS) - DLPFC/M1

INTERVENTIONS:
Device: Repetitive transcranial magnetic stimulation (rTMS) - M1/DLPFC — Repetitive transcranial magnetic stimulation (rTMS) is a treatment technique involving the induction of an electrical current on the surface of the cortex by applying a magnetic field to the scalp. This field is generated using a stimulation loop controlled by a robotic arm linked to a neuronavigation system. rTMS of M1 then rTMS of DLPFC.
  Other Names: rTMS
  Arms: M1 - DLPFC
Device: Repetitive transcranial magnetic stimulation (rTMS) - DLPFC/M1 — Repetitive transcranial magnetic stimulation (rTMS) is a treatment technique involving the induction of an electrical current on the surface of the cortex by applying a magnetic field to the scalp. This field is generated using a stimulation loop controlled by a robotic arm linked to a neuronavigation system. rTMS of DLPFC then rTMS of M1.
  Other Names: rTMS
  Arms: DLPFC - M1

SUMMARY:
High-frequency repetitive transcranial magnetic stimulation of the primary motor cortex has shown its effect on refractory neuropathic pain, and rTMS of the dorsolateral prefrontal cortex is commonly used for treatment-resistant depression.

The treatment for patients suffering from neuropathic pain and depression, concomitantly, still needs to be studied, as there are some specificities in both symptoms and brain functional MRI.

DETAILED DESCRIPTION:
This project is a cross-over study for these patients, including 4 sessions of either M1 or DLPFC rTMS, a wash-out period, followed by 4 sessions of the other stimulation site, to assess the efficiency of a DLPFC rTMS for neuropathic pain with a comorbid depression. Besides pain intensity and quality, patient's mood, quality of life, and catastrophizing will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Central or peripheral neuropathic pain
* Chronic pain (present for more than 6 months) with intensity greater than or equal to 4/10 on the numerical scale
* Pain present on a daily or near-daily basis (at least 4 days a week)
* Patient not completely relieved by recommended drug treatments for first- and second-line neuropathic pain
* Stable analgesic treatment (no new treatment or dosage adjustment) for at least one month, and will not need to be modified for the duration of the study.
* Patient with a depressive episode characterized according to DSM V criteria
* Indication for motor cortex rTMS by a neurologist
* Patient can be followed for the entire duration of the study
* Patient having received informed consent to participate in the study, and having co-signed a consent form with the investigator
* Member or beneficiary of a social security scheme

Exclusion Criteria:

* Industrial accident or litigation
* Contraindication to rTMS or MRI (seismotherapy treatment since the previous month; epilepsy and/or history of epilepsy; history of head trauma; neurosurgical lesion; intracranial hypertension; intracerebral metal clip; piercing; pacemaker; insulin pump; metal prosthesis; pregnant or breast-feeding woman; claustrophobia)
* Drug or psychoactive substance abuse
* Neuropathic pain in the context of a progressive pathology (HIV, cancer, systemic disease disease)
* Presence of other pain more severe than that justifying inclusion
* Patient unable to understand informed consent
* Patient unwilling or unable to stop treatments prohibited during the study
* Patient participating in another research protocol involving a drug within the 30 days prior to inclusion
* Patient deprived of liberty or under legal protection (guardianship, curatorship, safeguard of justice safeguard, family safeguard)
* Minor patient

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-26 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Comparison of pain relief rates between the two stimulation targets (M1 and DLPFC) | 2 weeks after the last rTMS session for each arm
  Patients are asked how much pain relief they have experienced since the last session.

SECONDARY OUTCOMES:
Neuropathic dimension | Up to 26 weeks
  Neuropathic dimension: overall score of the Neuropathic Pain Symptoms Inventory (NPSI) questionnaire and its dominant sub-score. The dominant being defined as the score of the dimension (e.g. allodynia, burning, dysesthesia) most painful at the inclusion visit (S0).This questionnaire is used to assess the presence and evolution of neuropathic pain symptoms, as well as the effectiveness of specific neuropathic pain treatments. Based on questioning, it comprises 12 questions (10 descriptive of symptoms and and 2 to assess pain frequency and duration).
  Score is from 0 ((no pain) to 120 (maximun pain)
Pain evolution | Up to 26 weeks
  Pain evolution via multiple Visual Analogue Scale (components: intensity, unpleasantness, impact on on attention). (Minimum Value : 0 means "no pain" - Maximum value : 10 means "the most intense pain imaginable").
Progression of depression (Montgomery Asberg Depression Rating Scale - MADRS) | 2 weeks after rTMS sessions
  Progression of depression (thymia), assessed by subjective percentage improvement in mood by the MADRS. Montgomery Asberg Depression Rating Scale (MADRS) consists of 10 items to be completed during a clinical interview. Each item has a severity scale from 0 to 6, with higher scores reflecting more severe symptoms. Scores can be added together to give an overall score (from 0 to 60).
Progression of depression (Beck Depression Inventory - BDI) | 2 weeks after rTMS sessions
  Progression of depression (thymia), assessed by subjective percentage improvement in mood by the Beck Depression Inventory (BDI). It provides a quantitative estimate of depression intensity. Each item consists of 4 sentences corresponding to 4 degrees of increasing intensity on a scale from 0 to 3. The overall score for the depressive syndrome (from 0 to 39) is obtained by adding up the scores for the 13 items.
Changes in mean pain intensity | 2 weeks after rTMS sessions
  Comparison of changes in mean pain intensity between the two treatment arms by using Visual Analogue Scale (components: intensity, unpleasantness, impact on on attention). (Minimum Value : 0 means "no pain" - Maximum value : 10 means "the most intense pain imaginable").
Evolution of catastrophism | 2 weeks after rTMS sessions
  Evolution of catastrophism via the Pain Catastrophizing Scale. People are asked to indicate the degree to which they have the above thoughts and feelings when they are experiencing pain using the 0 (not at all) to 4 (all the time) scale. A total score is yielded (ranging from 0-52), along with three subscale scores assessing rumination, magnification and helplessness.
Evolution of affective and sensory components of pain | 2 weeks after rTMS sessions
  Evolution of affective and sensory components of pain via the Pain Questionnaire Saint-Antoine (QDSA). This questionnaire contains 58 words divided into 16 categories offering dimensions that to describe the painful experience
Change in perceived quality of life | 2 weeks after rTMS sessions
  Change in perceived quality of life using the EuroQol-5D (EQ5-D). The answers given to ED-5D permit to find 243 unique health states or can be converted into EQ-5D index an utility scores anchored at 0 for death and 1 for perfect health. The EQ-5D questionnaire also includes a Visual Analog Scale (VAS), by which respondents can report their perceived health status with a grade ranging from 0 (the worst possible health status) to 100 (the best possible health status).
Adverse events | Up to 26 weeks
  Potential adverse events reporting during the study

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Saint-Etienne, Saint-Etienne, France